CLINICAL TRIAL: NCT02421289
Title: Influence of Cytochrome P2B6 on Efavirenz Dose in HIV-infected Thai Patients in a Prospective Randomized Controlled Trial: a Proof-of-concept Study
Brief Title: Influence of Cytochrome P2B6 on Efavirenz Dose in HIV-infected Thai Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Pansachee DAMRONGLERD, Ramathibodi Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID 05-56-13
Record Dates: First submitted 2015-04-08; First posted 2015-04-20 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Cytochrome P-450 CYP2B6; Efavirenz; HIV
Keywords: CYP2B6 polymorphism; efavirenz; Thai; HIV-infected patient; pharmacogenomic
MeSH Terms: interventions — efavirenz

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CYP2B6 guided group (Experimental): Patients were assigned to perform CYP2B6 study before ART initiation. If CYP2B6 *6/*6 was found in CYP2B6 *6/*6, the patients will be initiated a low dose of 400 mg of efavirenz (2 tablets of 200 mg) with tenofovir 300 mg and lamivudine 300 mg.
  Interventions: Drug: Efavirenz; Other: CYP450 2B6
- control group (No Intervention): Patients were promptly ART initiation regardless CYP2B6 results. Treatments were efvirenz 600 mg, tenofovir 300 mg and lamivudine 300 mg.

INTERVENTIONS:
Drug: Efavirenz — There will be adjusted dose of efavirenz in CYP2B6 guide group
  Arms: CYP2B6 guided group
Drug: Efavirenz — If the patients was diagnosed as hypersensitivity to EFV, they will receive boosted-PI instead.
  Arms: CYP2B6 guided group
Other: CYP450 2B6 — All patients will be monitored drug level which should be in therapeutic level.
  Arms: CYP2B6 guided group

SUMMARY:
Genetic polymorphisms of cytochrome P450 2B6 (CYP2B6) are associated with lower rate of EFV metabolism and lead to high exposure, as well as a higher risk of neuropsychiatric adverse event especially homozygous variant CYP2B6 *6/*6. This trial was designed to compare the proportion of patients who had undetectable HIV RNA at 24 weeks after ART initiation between patient who did CYP 2B6 guided EFV dose and who did not.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Anti-HIV positive
* Naïve to antiretroviral drugs
* Meet the criteria to start ART to Thai National guidelines
* Sign inform consent

Exclusion Criteria:

* Body mass index (BMI) >25 kg/m²
* Pregnant women or breastfeeding
* Received drugs that may have interaction with EFV e.g. rifampicin, fluconazole (400-800 mg), ergot alkaloid, midazolam, triazolam, ritonavir, carbamazepine, phenytoin, phenobarbitone, St John's Wort
* Having active opportunistic infections e.g. tuberculosis, cryptococcosis, histoplasmosis, penicillosis
* Hepatic dysfunction as indicated by:
* Transaminases >5-10 × the upper limit of normal
* ALP >5-10 × the upper limit of normal
* Total bilirubin >2.5-5 × the upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
HIV RNA | 24 weeks

SECONDARY OUTCOMES:
Neuropsychiatric adverse events | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pansachee Damronglerd, M.D., Principal Investigator — Faculty of medicine Ramathibodi Hospital
Locations (1):
- Faculty of medicine Ramathibodi Hospital, Bangkok, Bangkok, Thailand